CLINICAL TRIAL: NCT02367001
Title: Randomized Trial Evaluating the Effectiveness of a "Targeted Communication" With the General Practitioner Involvement in Cancer Screening Invitation Letters
Brief Title: Randomized Trial Evaluating the Effectiveness of the General Practitioner Involvement in Cancer Screening Invitations
Acronym: GPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: INCA-P3644-KH-GPs
Record Dates: First submitted 2015-01-28; First posted 2015-02-20 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Cervical Cancer
Keywords: general practitioner; screening; participation; organized screening
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: standard invitation (Other): Group 1: sending a standard invitation signed by the coordinating doctor (send by the structure responsible for organized screenings)
  Intervention : Normal invitation
  Interventions: Other: Normal invitation
- 2: Revised invitation (Experimental): Group 2: Sending a revised invitation ( text, layout) signed by the coordinating doctor (send by the structure responsible for organized screenings)
  Intervention : revised invitation signed by the coordinating doctor
  Interventions: Other: revised invitation signed by the coordinating doctor
- 3 : revised invitation signed by the attending physician (Experimental): Group 3: Sending a revised invitation signed by the attending physician (send by the structure responsible for organized screenings)
  Intervention : Revised invitation signed by the attending physician
  Interventions: Other: Revised invitation signed by the attending physician

INTERVENTIONS:
Other: Normal invitation — No modification and signed by the coordinating doctor as usual
  Arms: 1: standard invitation
Other: revised invitation signed by the coordinating doctor — Invitation with revised text and layout and signed by the coordinating doctor as usual
  Arms: 2: Revised invitation
Other: Revised invitation signed by the attending physician — signature typed or typed + handwritten
  Arms: 3 : revised invitation signed by the attending physician

SUMMARY:
Our goal is to evaluate, in France, the effectiveness (in terms of participation) of the general practitioner involvement (signature) and a more personalized communication in invitation letters to organized screening of breast, colorectal and cervical cancers.

The hypothesis on which this project is based is that communication is probably more effective if the "receiver" feels personally targeted by invitation letters (Dear Martin, I am writing ...) and if he knows "the issuer "(his general practitioner rather an unknown person).

ELIGIBILITY:
Inclusion Criteria:

* Living in Indre-et-Loire (french territorial division 37)
* Be affiliated to the following three health insurance companies: CPAM (Caisse Primaire d'Assurance Maladie), MSA (Mutualité Sociale Agricole), or RSI (Régime social des Indépendants)
* Having declared (to health insurance company) an attending physician who has given its written consent to participate in the study
* Present no exclusion criterion to cancer screening ( for each one)
* Be old from 50 to 74 years (breast and colorectal cancer) or from 25 to 65 years (cervical cancer)

Exclusion Criteria:

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53978 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect on the participation (of the population) in cancer screening of an intervention involving the general practitioner (integration of signature) in the invitation letters | 9 or 12 months after the invitation letters
  The participation / non participation will be measured for each cancer screening (breast, colorectal and cervical) :
  * 9 months after the invitation letters for breast and colorectal cancers
  * 12 months after the invitation letters for cervical cancer
  The participation rate is defined as the number of people having participated, divided by the total number of people in the group or subgroup considered.
  Analysis by comparing the participation rates between groups (Group 1, Group 2 and Group 3) and sub-groups will be done.

SECONDARY OUTCOMES:
Evaluate the effectiveness on the participation (of the population) of the use of a simplified and more focused communication in the invitation letters : comparison of the participation rates in arm 1 (normal invitation) and arm 2 (revised invitation) | 9 or 12 months after the invitation letters
Evaluate the effectiveness on the participation (of the population) of the two types of general practitioner signature (typed versus typed + handwritten) by comparing the participation rates between two sub-groups in the arm 3. | 9 or 12 months after the invitation letters
Cost-effectiveness of different strategies for each cancer screening (breast, colorectal and cervical) as measured by cost effectiveness ratio (total costs in Euros divided by total screened people) | 9 or 12 months after the invitation letters

CONTACTS AND LOCATIONS:
Overall Officials: Ken HAGUENOER, Study Director — University Hospital of TOURS
Locations (1):
- Centre de Coordination des Dépistages des Cancers (CCDC), Tours, France